CLINICAL TRIAL: NCT05502471
Title: Serum Occludin and Zonulin Levels in Attention-deficit/Hyperactivity Disorder
Brief Title: Occludin and Zonulin in Attention-deficit/Hyperactivity Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Hicran Dogru, MD, Ataturk University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 025
Record Dates: First submitted 2022-08-13; First posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Attention-deficit/Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADHD (Other): Children with ADHD
  Interventions: Diagnostic Test: Zonulin; Diagnostic Test: Occludin
- Control (Other): Children without any psychiatric disorder
  Interventions: Diagnostic Test: Zonulin; Diagnostic Test: Occludin

INTERVENTIONS:
Diagnostic Test: Zonulin — Serum zonulin level
Diagnostic Test: Occludin — Serum occludin level

SUMMARY:
The association between levels of zonulin and occludin and behavioral/emotional problems in children with ADHD are investigated.

DETAILED DESCRIPTION:
Inclusion criteria for the ADHD group are (a) newly diagnosed ADHD (b) no prior psychotropic treatment for ADHD or any psychiatric disorder (c) age 6-12 years. Exclusion criteria were: (a) history of history of inflammatory/noninflammatory, metabolic, or autoimmune disease (b) any special diet history within the past year (c) use of corticosteroids or regular intake of medication in the last 6 months, (d) body mass index (BMI) [kg/m2] > 30), and (e) cognitive deficits by developmental history.

ELIGIBILITY:
Inclusion Criteria:

* (a) newly diagnosed ADHD
* (b) no prior psychotropic treatment for ADHD or any psychiatric disorder
* (c) age 6-12 years.

Exclusion Criteria:

* (a) history of history of inflammatory/noninflammatory, metabolic, or autoimmune disease
* (b) any special diet history within the past year
* (c) use of corticosteroids or regular intake of medication in the last 6 months,
* (d) body mass index (BMI) [kg/m2] > 30),
* (e) cognitive deficits by developmental history

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 79 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Zonulin level | 1 month
  Serum Zonulin level after psychiatric interview
Occludin level | 1 month
  Serum Occludin level after psychiatric interview

CONTACTS AND LOCATIONS:
Overall Officials: Hicran Dogru, MD, Principal Investigator — Ataturk University
Locations (1):
- Ataturk University Hospital, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No